CLINICAL TRIAL: NCT07370129
Title: Impact of Transnasal Sphenopalatine Ganglion Block on Pain Relief and Recovery Following Tonsillectomy
Brief Title: Transnasal Sphenopalatine Ganglion Block for Postoperative Pain and Recovery in Tonsillectomy (TONwoPA)
Acronym: TONwoPA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Sıddık Aytuğ, MD Sıddık Aytuğ Medical Resident, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025000458; 25-AKD-116 (Registry Identifier: Turkish Medicines and Medical Devices Agency)
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Post Tonsillectomy Pain; Post Operative Analgesia; Opioid Consumption; Sphenopalatine Ganglion Block; Tonsillar Surgery Complications
Keywords: Transmucosal Sphenopalatine Ganglion Block; Sphenopalatine Ganglion Block; Tonsillectomy Without Pain
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled interventional clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Lidocain (Experimental): Transnasal sphenopalatine ganglion block will be performed using cotton-tipped applicators soaked with 5% lidocaine hydrochloride, which will be prepared by diluting 10% lidocaine hydrochloride with 0.9% sodium chloride (normal saline).
  Interventions: Procedure: Transnasal Transmucosal Sphenopalatine Ganglion Block; Procedure: Lidocaine %5
- Group Saline (Sham Comparator): In the comparison group, a transnasal sphenopalatine ganglion block will be performed as a placebo using cotton-tipped applicators soaked with 0.9% sodium chloride (normal saline).
  Interventions: Procedure: Transnasal Transmucosal Sphenopalatine Ganglion Block; Procedure: Saline (0.9% NaCl)

INTERVENTIONS:
Procedure: Transnasal Transmucosal Sphenopalatine Ganglion Block — Before the start of surgery, a preemptive transnasal transmucosal sphenopalatine ganglion block will be performed using cotton-tipped applicators. The assigned solutions will be administered via the applicators according to group allocation.
Procedure: Lidocaine %5 — Transnasal Transmucosal Sphenopalatine Ganglion Block with Lidocaine %5
  Arms: Group Lidocain
Procedure: Saline (0.9% NaCl) — Transnasal Transmucosal Sphenopalatine Ganglion Block with Saline (0.9% NaCl)
  Arms: Group Saline

SUMMARY:
The aim of this clinical trial is to evaluate the effectiveness of transnasal transmucosal sphenopalatine ganglion block in reducing post-tonsillectomy pain. The study also investigates its impact on rescue analgesic requirements and postoperative recovery by comparing 5% lidocaine with placebo.

Participants will receive a transnasal transmucosal sphenopalatine ganglion block with either 5% lidocaine or placebo (saline). Postoperative pain levels and opioid consumption will be monitored during the first 24 hours after surgery. In addition, length of hospital stay, the occurrence of primary and secondary post-tonsillectomy hemorrhage up to 14 days, unplanned hospital readmissions after discharge, and patient satisfaction on postoperative day 14 will be assessed.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effects of preemptive transnasal transmucosal sphenopalatine ganglion block performed with either 0.9% saline (placebo) or 5% lidocaine (active drug), in addition to standard multimodal analgesia, on postoperative pain and recovery in patients aged 12 years and older undergoing tonsillectomy.

All patients will undergo routine monitoring, including noninvasive blood pressure, electrocardiography (ECG), peripheral oxygen saturation (SpO₂), body temperature, end-tidal carbon dioxide (ETCO₂), and bispectral index (BIS), followed by induction of general anesthesia.

For induction of general anesthesia, intravenous lidocaine 1 mg/kg, fentanyl 1 µg/kg, and propofol 1-3 mg/kg (adjusted according to depth of anesthesia monitoring) will be administered. Neuromuscular blockade required for endotracheal intubation and surgery will be achieved with intravenous rocuronium 0.8 mg/kg. Airway security will be ensured by orotracheal intubation. Anesthesia maintenance will be provided as total intravenous anesthesia (TIVA) using a propofol and remifentanil combination, guided by BIS monitoring.

Immediately after induction of anesthesia, patients will be randomized into either the Saline Group (placebo) or the Lidocaine Group (5% lidocaine, active drug) using a computer-generated randomization program.

Before the start of surgery, a preemptive transnasal transmucosal sphenopalatine ganglion block will be performed. Patients in the placebo group will receive 0.9% isotonic saline, while patients in the lidocaine group will receive 5% lidocaine. Cotton-tipped applicators will be used for the block procedure, with one applicator inserted into each nostril. The applicators will be advanced parallel to the nasal floor from the middle turbinate until resistance is encountered. Contact of the applicator with the posterior wall of the nasopharynx will ensure transmucosal proximity to the sphenopalatine ganglion. The assigned solutions will be applied via the applicators according to group allocation, aiming for transmucosal absorption and therapeutic effect on the target ganglion.

The applicators will be shortened as necessary to avoid interference with the surgical field and will be left in place throughout the surgery. Before emergence from anesthesia, the same solution will be reapplied through the applicators. Patients will be awakened approximately 10 minutes after the second application, prior to extubation. The total volume of solution administered per patient will be 3 mL: 2 mL (1 mL per applicator) before surgery and 1 mL (0.5 mL per applicator) after surgery.

As part of standard multimodal analgesia, all patients will receive intravenous paracetamol 1 g, ibuprofen 400 mg, and dexamethasone 8 mg. For postoperative nausea and vomiting prophylaxis, ondansetron 4 mg IV will be administered before the end of surgery. Extubation will be performed after neuromuscular recovery is confirmed with a train-of-four (TOF) ratio ≥ 0.9, using sugammadex as needed.

Following transfer to the post-anesthesia care unit (PACU), all patients will receive intravenous fentanyl via patient-controlled analgesia (PCA) and will continue to be monitored using standardized case report forms. Fentanyl PCA will be prepared for all patients with a concentration of 10 µg/mL, a bolus dose of 0.2 µg/kg, a lockout interval of 12 minutes, and a maximum dose of 5 µg/kg over a 4-hour period.

In the preoperative period, demographic data of all patients will be recorded along with American Society of Anesthesiologists (ASA) physical status, Mallampati score, and Brodsky Tonsil Hypertrophy Scale. The presence of preoperative dysphagia, aspiration risk, and throat pain will also be documented.

During the intraoperative period, whether endotracheal intubation is achieved on the first attempt and the occurrence of any complications during intubation or extubation (including the type of complication, if present) will be recorded. In addition, heart rate (HR), arterial blood pressure values (systolic, diastolic, and mean arterial pressure [MAP]), peripheral oxygen saturation (SpO₂), end-tidal carbon dioxide (ETCO₂), and bispectral index (BIS) values will be recorded before anesthesia induction, after induction (corresponding to the pre-block period), and every 5 minutes intraoperatively.

Postoperative follow-up will be performed in the post-anesthesia care unit (PACU), at postoperative hours 1, 2, 4, 8, 16, and 24, and on postoperative day 14. In the PACU, patients will be evaluated by an anesthesiologist for pain (assessed using the Numeric Rating Scale [NRS]), postoperative nausea and vomiting, and potential airway-related complications, including aspiration, hoarseness, laryngospasm, dyspnea, stridor, and oxygen requirement. Patients with a Modified Aldrete Score ≥ 9 will be discharged from the PACU.

At postoperative hours 1, 2, 4, 8, 16, and 24, NRS pain scores will be recorded. In addition, the presence of nausea and vomiting, the need for additional (rescue) analgesia, and any airway-related complications will be documented. The time to first oral intake of fluids and solid foods, as well as any associated pain during oral intake, will also be monitored.

Finally, length of hospital stay, the occurrence of primary and secondary post-tonsillectomy hemorrhage up to postoperative day 14, any unplanned hospital readmissions after discharge, and patient satisfaction on postoperative day 14 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 12 years
* Patients weighing ≥ 50 kg
* Patients without coagulation disorders
* ASA physical status I-II patients scheduled for tonsillectomy
* Patients who are fully oriented and able to cooperate

Exclusion Criteria:

* Lack of informed consent
* Patients aged < 12 years
* Patients weighing < 50 kg
* Body mass index (BMI) > 30 kg/m²
* History of allergy to local anesthetics
* History of facial trauma or infection
* Presence of coagulation disorders
* Patients who are disoriented and/or unable to cooperate
* Patients with comorbidities requiring opioid use
* History of neuropathic pain
* Patients with chronic pain syndrome

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative NRS Score and Opioid Consumption | Postoperative 1. 2. 4. 8. 16. and 24. Hours
  The NRS (Numeric Rating Scale) score will be used to assess the pain during follow ups. Scale: 0 (no pain) to 10 (worst pain). Higher scores on the NRS indicate worse pain.

SECONDARY OUTCOMES:
Parameters for Postoperative Complications and Recovery Process | Postoperative 14th Day
  Length of hospital stay, the occurrence of primary and secondary post-tonsillectomy hemorrhage up to postoperative day 14, the presence of any complaints requiring unplanned hospital readmission after discharge, and patient satisfaction on postoperative day 14 will be assessed.
Feeding Tolerance and Time to First Tolerated Oral Intake | Postoperative 1.2.4.8.16. and 24. Hours
  The timing of the patient's first oral intake of liquids and solids, and any accompanying pain, will also be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Aşık, Professor, Study Chair — Ankara University
Locations (1):
- Ankara University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study was not designed with a data-sharing plan and to ensure participant confidentiality.

REFERENCES:
- [Background] Nelson Textbook of Pediatrics Twenty Second Edition Pediatric Pain Management Nelson Textbook of Pediatrics, Chapter 93, 677-700.e2
- [Background] Rajan S, Sasikumar NK, Rudrahitlu V, Mathew J, Barua K, Kumar L. Effects of bilateral transmucosal sphenopalatine ganglion block on intraoperative anesthetic requirements and recovery profile in children undergoing palatoplasty under general anesthesia. J Anaesthesiol Clin Pharmacol. 2023 Apr-Jun;39(2):220-225. doi: 10.4103/joacp.joacp_279_21. Epub 2023 Feb 3. PMID 37564832
- [Background] Sphenopalatine ganglion block for the treatment of postdural puncture headache: a randomised, blinded, clinical trial British Journal of Anaesthesia, 124 (6): 739e747 (2020) doi: 10.1016/j.bja.2020.02.025
- [Background] Bucard BM, Assad AR, Vercosa N, Cavalcanti IL. Sphenopalatine ganglion block for postoperative analgesia after transsphenoidal hypophysectomy: A pilot study. Eur J Anaesthesiol. 2025 Apr 1;42(4):368-370. doi: 10.1097/EJA.0000000000002112. Epub 2025 Jan 9. No abstract available. PMID 39789934
- [Background] Rezaeian A, Hashemi SM, Dokhanchi ZS. Effect of Sphenopalatine Ganglion Block With Bupivacaine on Postoperative Pain in Patients Undergoing Endoscopic Sinus Surgery. Allergy Rhinol (Providence). 2019 Jan 23;10:2152656718821282. doi: 10.1177/2152656718821282. eCollection 2019 Jan-Dec. PMID 30719401
- [Background] Piagkou M, Demesticha T, Troupis T, Vlasis K, Skandalakis P, Makri A, Mazarakis A, Lappas D, Piagkos G, Johnson EO. The pterygopalatine ganglion and its role in various pain syndromes: from anatomy to clinical practice. Pain Pract. 2012 Jun;12(5):399-412. doi: 10.1111/j.1533-2500.2011.00507.x. Epub 2011 Sep 29. PMID 21956040
- [Background] Robbins MS, Robertson CE, Kaplan E, Ailani J, Charleston L 4th, Kuruvilla D, Blumenfeld A, Berliner R, Rosen NL, Duarte R, Vidwan J, Halker RB, Gill N, Ashkenazi A. The Sphenopalatine Ganglion: Anatomy, Pathophysiology, and Therapeutic Targeting in Headache. Headache. 2016 Feb;56(2):240-58. doi: 10.1111/head.12729. Epub 2015 Nov 30. PMID 26615983
- [Background] Smith L, Balakrishnan K, Pan S, Tsui BCH. Suprazygomatic maxillary (SZM) nerve blocks for perioperative pain control in pediatric tonsillectomy and adenoidectomy. J Clin Anesth. 2021 Aug;71:110240. doi: 10.1016/j.jclinane.2021.110240. Epub 2021 Mar 20. No abstract available. PMID 33756446
- [Background] Mahrose R, Shorbagy MS, Kasem AA. Opioid Free Ptyregopalatine Ganglion Block Based Multimodal Anesthesia Versus Conventional Opioid Based Multimodal Anesthesia for Tonsillectomy Operations: A Randomized Controlled Trial. Anesth Pain Med. 2024 Jul 10;14(3):e146617. doi: 10.5812/aapm-146617. eCollection 2024 Jun. PMID 39416797
- [Background] Vlok R, Melhuish TM, Chong C, Ryan T, White LD. Adjuncts to local anaesthetics in tonsillectomy: a systematic review and meta-analysis. J Anesth. 2017 Aug;31(4):608-616. doi: 10.1007/s00540-017-2310-x. Epub 2017 Jan 24. PMID 28120104
- [Background] Ahmed SA, Omara AF. The Effect of Glossopharyngeal Nerve Block on Post-Tonsillectomy Pain of Children; Randomized Controlled Trial. Anesth Pain Med. 2019 Apr 30;9(2):e90854. doi: 10.5812/aapm.90854. eCollection 2019 Apr. PMID 31341828
- [Background] Park HP, Hwang JW, Park SH, Jeon YT, Bahk JH, Oh YS. The effects of glossopharyngeal nerve block on postoperative pain relief after tonsillectomy: the importance of the extent of obtunded gag reflex as a clinical indicator. Anesth Analg. 2007 Jul;105(1):267-71. doi: 10.1213/01.ane.0000266440.62424.f1. PMID 17578986
- [Background] Mohamed SK, Ibraheem AS, Abdelraheem MG. Preoperative intravenous dexamethasone combined with glossopharyngeal nerve block: role in pediatric postoperative analgesia following tonsillectomy. Eur Arch Otorhinolaryngol. 2009 Nov;266(11):1815-9. doi: 10.1007/s00405-009-0937-4. Epub 2009 Mar 5. PMID 19263066
- [Background] Fedorowicz Z, van Zuuren EJ, Nasser M, Carter B, Al Langawi JH. Oral rinses, mouthwashes and sprays for improving recovery following tonsillectomy. Cochrane Database Syst Rev. 2013 Sep 10;2013(9):CD007806. doi: 10.1002/14651858.CD007806.pub4. PMID 24022333
- [Background] Bean-Lijewski JD. Glossopharyngeal nerve block for pain relief after pediatric tonsillectomy: retrospective analysis and two cases of life-threatening upper airway obstruction from an interrupted trial. Anesth Analg. 1997 Jun;84(6):1232-8. doi: 10.1097/00000539-199706000-00011. PMID 9174298
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387
- [Background] Colvin LA, Bull F, Hales TG. Perioperative opioid analgesia-when is enough too much? A review of opioid-induced tolerance and hyperalgesia. Lancet. 2019 Apr 13;393(10180):1558-1568. doi: 10.1016/S0140-6736(19)30430-1. PMID 30983591
- [Background] Nafziger AN, Barkin RL. Opioid Therapy in Acute and Chronic Pain. J Clin Pharmacol. 2018 Sep;58(9):1111-1122. doi: 10.1002/jcph.1276. Epub 2018 Jul 9. PMID 29985526
- [Background] Smith CR, Helander E, Chheda NN. Trigeminal Nerve Blockade in the Pterygopalatine Fossa for the Management of Postoperative Pain in Three Adults Undergoing Tonsillectomy: A Proof-of-Concept Report. Pain Med. 2020 Oct 1;21(10):2441-2446. doi: 10.1093/pm/pnaa062. PMID 32232479
- [Background] Ozkiris M, Kapusuz Z, Saydam L. Comparison of three techniques in adult tonsillectomy. Eur Arch Otorhinolaryngol. 2013 Mar;270(3):1143-7. doi: 10.1007/s00405-012-2160-y. Epub 2012 Aug 22. PMID 23010796
- [Background] Paganelli A, Ayari Khalfallah S, Brunaud A, Constant I, Deramoudt V, Fayoux P, Giovanni A, Mareau C, Marianowski R, Michel J, Mondain M, Schultz P, Treluyer JM, Wood C, Pondaven S, Nicollas R; SFORL Work Group. Guidelines (short version) of the French Oto-Rhino-Laryngology--Head and Neck Surgery Society (SFORL) for the management of post-tonsillectomy pain in adults. Eur Ann Otorhinolaryngol Head Neck Dis. 2014 Sep;131(4):227-32. doi: 10.1016/j.anorl.2014.05.003. Epub 2014 Aug 5. PMID 25106699
- [Background] Ericsson E, Brattwall M, Lundeberg S. Swedish guidelines for the treatment of pain in tonsil surgery in pediatric patients up to 18 years. Int J Pediatr Otorhinolaryngol. 2015 Apr;79(4):443-50. doi: 10.1016/j.ijporl.2015.01.016. Epub 2015 Jan 24. PMID 25677565
- [Background] Persino PR, Saleh L, Walner DL. Pain control following tonsillectomy in children: A survey of patients. Int J Pediatr Otorhinolaryngol. 2017 Dec;103:76-79. doi: 10.1016/j.ijporl.2017.10.016. Epub 2017 Oct 7. PMID 29224770
- [Background] Aldamluji N, Burgess A, Pogatzki-Zahn E, Raeder J, Beloeil H; PROSPECT Working Group collaborators*. PROSPECT guideline for tonsillectomy: systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Jul;76(7):947-961. doi: 10.1111/anae.15299. Epub 2020 Nov 17. PMID 33201518
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Darrow DH, Siemens C. Indications for tonsillectomy and adenoidectomy. Laryngoscope. 2002 Aug;112(8 Pt 2 Suppl 100):6-10. doi: 10.1002/lary.5541121404. PMID 12172229